CLINICAL TRIAL: NCT05273398
Title: Exploratory Open-Label Study of Effects on Responsive Neurostimulator Activity After Intranasal Administration of Single Dose of Valtoco® to People With Epilepsy
Brief Title: Effects of Diazepam on RNS Detections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael Privitera, Professor Neurology, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0017
Record Dates: First submitted 2022-02-17; First posted 2022-03-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Epilepsies, Partial
Keywords: epilepsy; responsive neurostimulator; diazepam; rescue medication
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Diazepam

STUDY DESIGN:
Intervention Model Description: 4 subject pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Single arm of treatment
  Interventions: Drug: nasal diazepam

INTERVENTIONS:
Drug: nasal diazepam — Nasal administration of diazepam
  Other Names: Nasal diazepam (Valtoco)

SUMMARY:
To assess the magnitude and duration of reduction in RNS recorded Detections and Long Episodes following intranasal administration of Valtoco®. All participants will have been implanted and treated with an RNS system for clinical purposes and regularly upload Detection and Long Episode data on a regular basis as part of regular clinical treatment. Participants will come to the clinic and be administered a single dose of Valtoco® via nasal spray. RNS recorded Detections and Long Episodes before and after Valtoco® administration will be compared. This is a pilot study, so all outcomes are exploratory.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the impact of Valtoco® administration on events recorded by RNS compared to the same time administration of the prior seven days.

Objectives: The investigators will assess the percent change in Detections calculated separately for each hour during the first 8 hours of the post-dose observation period. The number of Detections during each hour of the 8-hour period post dose will be compared to the same hour during the seven comparable 8-hour sessions of the 7-day pre-dose observation period. That is, if the dose was given at 9 AM on day 0, then the mean number of Detections at baseline will be calculated as the mean number of Detections from 9 AM to 10 AM on day -1 through day -7. The percent change in Detections will be calculated as (number of Detections in hour 1 post dose)/(Mean number of Detections in hour 1 on Day -1 through Day -7). The same hourly change will be calculated for each of the 8 hours after dosing. The comparison will be the same hours each day to minimize the hour to hour variability typically seen in these measures.

Hourly histograms generated by the RNS system and stored in the PDMS will be collected. In addition, using "detailed diagnostics" visual analysis of minute-by-minute Detections will be reviewed for obvious patterns of interest for the 8 hours post dosing.

Total number of hours during the 48-hour post-dose observation period where the number of Detections is <50% of the mean hourly Detection rate over the 7-day pre-dose observation period will be calculated.

The number of Long Episodes recorded during the 7-day pre-dose observation period will be compared to the number of Long Episodes during the post-dose 48-hour observation period.

The number of diary-recorded seizures during the post-dose observation period will be recorded.

The investigators will quantify the 2 highest hourly detection rates for the 7-day pre-dose and 48-hour post-dose periods.

The investigators will calculate the number of days required for the daily detection rate to fall within the 90% confidence interval of the 9 am to 5 PM baselines from the 7-day pre-dose baseline.

The investigators will use descriptive statistics for the detection data and Long Episodes for the entire 7-day post dose period.

The investigators will quantify the time course of observable changes in beta activity on the ECoG recorded samples on the day of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria (participants must meet all Inclusion Criteria)

  1. Age 18 or above
  2. Participant will weigh >50 Kg.
  3. RNS will have been implanted for usual treatment for at least 3 months. Detection settings will be stable at least 30 days.
  4. No changes in AED dosages, VNS settings (if participant has VNS) or RNS detection or stimulation parameters 30 days before and during the study. However, patients with newer VNS models that have tachycardia detection will be excluded because of the variability of the stimulations, which could affect RNS Detections. If the VNS device that uses tachycardia detection can be inactivated, the patient would not be excluded from participating in the study.
  5. Minimum mean rate of Detections of 5 (NUMBER CHANGED) per hour during the hours of 9 AM to 5 PM, and no fewer than 2 (NUMBER CHANGED) Detections in any hour between 9 AM and 5 PM in the pre-dose baseline observation period. Pre-dose baseline observation period will be 7 days in duration, from day -7 to day 0 prior to dosing.
  6. Participant must meet criteria for Detection variability based on historical Detections. No more than 97% (NUMBER CHANGED) change in highest to lowest hour detection during the 9 AM to 5 PM observation period OF A SINGLE DAY. Calculation will be (highest hourly detection rate - lowest hourly detection rate)/highest hourly detection rate= <0.97 (NUMBER CHANGED). For example: highest hourly detection rate = 1000; lowest hourly detection rate = 300, (1000-300)/1000 = 0.7, and this patient would meet qualifying criteria.
  7. If the participant fails the minimal mean Detection rate criteria or Detection variability criteria during the screening period, one additional screening period for RNS Detections may take place a minimum of one week later.
  8. If the participant fails screening due to a clinical seizure in the 96 hours prior to dosing, two additional screening periods for Detection and seizures may be undertaken.
  9. Focal epilepsy consistent with ILAE criteria supported by either EEG or MRI data and meets ILAE definition of refractory epilepsy.
  10. May be on stable prescribed dose of Selective Serotonin Reuptake Inhibitor (SSRI), Serotonin-Norepinephrine Reuptake Inhibitor (SNRI), or atypical antipsychotic for at least 3 months
  11. Optimal candidates will have temporal lobe RNS implantation, but extra-temporal implantation is acceptable if minimal Detection rate criteria are met.

Exclusion Criteria:

Exclusion:

1. Pregnancy; every woman of childbearing age will be asked at every visit, "Do you think that you might be pregnant?" If yes, a pregnancy test will be administered. Any woman with a positive test will be excluded from participation.
2. Not competent to sign consent
3. Any history of substance abuse within the previous 2 years.
4. Cannabidiol as EpidiolexR on a stable dose, will be the only allowed cannabinoid. Subjects with recreational or medicinal use of marijuana, cannabinoids and/or derivatives in the prior 30 days will be excluded.
5. Current chronic opioid use.
6. History of poor medication compliance as judged by the investigator
7. Any medical or psychiatric condition that the investigator believes would impair reliable participation in the trial
8. Subject is participating or has participated in an investigational product/device trial currently or in the preceding 30 days.
9. Subject has been diagnosed with only psychogenic or non-epileptic seizures.
10. Use of rescue benzodiazepines less than two weeks before baseline detection rate assessment begins. Stable doses of a prescribed benzodiazepine for 30 days prior to study entry is permitted.
11. Benzodiazepines used intermittently or on an as needed basis for sleep will not be allowed for the 7 days prior to and 7 days following the Valtoco dose.
12. No clinical seizure during the period starting 48 hours before pre-dose baseline observation period begins (i.e., 96 hours before dose is administered) until 48 hours after the Valtoco administration. If a clinical seizure occurs during the 48-hour pre-dose baseline period, the potential participant can be re-screened after one week. If a clinical seizure occurs within 8 hours of dosing, the participant may repeat screening and dose after one week. If a clinical seizure occurs more than 8 hours after dosing, the PI will assess whether the first 8-hour data is sufficient or whether a re-screening and dose should take place.
13. A history of allergy to diazepam or midazolam, or any of the ingredients of Valtoco®.
14. A history of adverse reaction to diazepam or midazolam that in the opinion of the investigator would jeopardize the health of the participant or interfere with interpretation of study results.
15. A history of narrow-angle glaucoma or inadequately treated open-angle glaucoma
16. Large variations in RNS detections that in the opinion of the investigator would interfere with the ability to detect a drug effect on detections. Examples may include, but are not limited to, clusters of detections lasting a few days in duration or a high degree of cyclic clusters of detections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Detections | 8 days
  The investigators will assess the percent change in Detections calculated separately for each hour during the first 8 hours of the post-dose observation period. The number of Detections during each hour of the 8-hour period post dose will be compared to the same hour during the seven comparable 8-hour sessions of the 7-day pre-dose observation period.

SECONDARY OUTCOMES:
Change in hourly histograms | 8 hours
  Hourly histograms generated by the RNS system and stored in the PDMS will be collected. In addition, using "detailed diagnostics" visual analysis of minute-by-minute Detections will be reviewed for obvious patterns of interest for the 8 hours post dosing.
Detection reduction of >50% | 9 days
  Total number of hours during the 48-hour post-dose observation period where the number of Detections is <50% of the mean hourly Detection rate over the 7-day pre-dose observation period will be calculated.
Change in diary recorded seizures | 14 days
  The number of diary-recorded seizures during the post-dose observation period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Privitera, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Detection rates before and after administration of intranasal diazepam will be made available.